CLINICAL TRIAL: NCT00512200
Title: Postoperative Cognitive Dysfunction in Geriatric Patients: the Role of Intraoperative Cerebral Perfusion and Perioperative Anticholinergic Medication
Brief Title: Postoperative Cognitive Dysfunction in Geriatric Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: EK 75/07
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Delirium, Dementia, Amnestic, Cognitive Disorders; Postoperative Complications; Memory Disorders
MeSH Terms: conditions — Neurocognitive Disorders; Postoperative Complications; Memory Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Case: Patients aged 65 or older
- Control: Patients aged 20 to 40
- Control 2: Healthy volunteers aged 65 or older

SUMMARY:
Geriatric patients have a high risk of developing postoperative cognitive deficits. Hypothetical causes are insufficient intraoperative cerebral perfusion or drugs that are administered in the perioperative setting. This study will investigate the role of these two factors in patients aged 65 or older undergoing elective surgical procedures under general aesthesia. Non-invasive techniques will be used to monitor intraoperative cerebral perfusion and anticholinergic activity in the patient's blood is determined. Data will be compared to those of a young (20-40 year old) group of patients undergoing elective surgical procedures using an identical anesthetic technique. A second control group of healthy volunteers older than 65 will be investigated to quantify practice effects with repeated testing of cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgical procedure under general anaesthesia

Exclusion Criteria:

* History of cerebrovascular disease
* Mini Mental status <23
* Cardiac surgery
* Neurosurgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients undergoing elective major surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2007-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function due to surgery under general aesthesia | cognitive function measured prior to and after surgery
  cognitive function measured by Consortium to Establish a Registry for Alzheimer's Disease (CERAD) neurological test battery

CONTACTS AND LOCATIONS:
Overall Officials: Luzius A Steiner, MD, Prof., Principal Investigator — Department of Anaesthesia, University Hospital Basel
Locations (1):
- Department of Anaesthesia, University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Goettel N, Patet C, Rossi A, Burkhart CS, Czosnyka M, Strebel SP, Steiner LA. Monitoring of cerebral blood flow autoregulation in adults undergoing sevoflurane anesthesia: a prospective cohort study of two age groups. J Clin Monit Comput. 2016 Jun;30(3):255-64. doi: 10.1007/s10877-015-9754-z. Epub 2015 Aug 19. PMID 26285741